CLINICAL TRIAL: NCT05859269
Title: Methylprednisolone Taper After Total Knee Replacement: A Prospective Randomized Trial
Brief Title: Methylprednisolone Taper After Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ajay Premkumar, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005985
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Knee Arthritis
Keywords: Methylprednisolone; Total Knee Replacement
MeSH Terms: interventions — Methylprednisolone; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: Medrol Dose (Experimental): The perioperative Medrol dose treatment will consist of a course that lasts six days, with 24 milligrams administered on the first day, 20 milligrams on the second day, 60 milligrams on the third day, 12 milligrams on the fourth day, 8 milligrams on the fifth day, and 4 milligrams on the sixth day. Patients will then be followed up at the clinic for six weeks following their procedure to allow for clinical evaluation and to measure outcome variables.
  Interventions: Drug: Methylprednisolone
- Control Group: Standard of Care (Active Comparator): Patients in this group will receive a single intraoperative dose of 10 mg intravenous dexamethasone (control group, IV dexamethasone is standard of care).
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Methylprednisolone — Patients will receive a single intraoperative dose of 10 mg intravenous dexamethasone followed with a 6-day oral methylprednisolone taper course.
  Patients will also receive a standardized multimodal postoperative pain management regimen which includes nonsteroidal anti-inflammatory medication (e.g., NSAIDs) and opioid pain medications, both in the hospital and at home as part of standard care.
  Arms: Experimental Group: Medrol Dose
Other: Standard of Care — Patients will receive a single intraoperative dose of 10 mg intravenous dexamethasone (control group, IV dexamethasone is standard of care).
  Patients will also receive a standardized multimodal postoperative pain management regimen which includes nonsteroidal anti-inflammatory medication (e.g., NSAIDs) and opioid pain medications, both in the hospital and at home as part of standard care.
  Arms: Control Group: Standard of Care

SUMMARY:
Total knee replacement surgery is a commonly performed and widely successful surgery to improve mobility and decrease pain in patients suffering from severe knee arthritis. However, in the immediate period after knee replacement, patients often experience significant pain and nausea, which can limit early recovery after surgery. Glucocorticoids are anti-inflammatory drugs that can reduce pain and swelling by blocking the inflammatory process, and have already shown promise in various surgical settings, including after knee replacement. There are different glucocorticoid formulations available, and in this particular study, we are evaluating the effects of administering a Medrol Dose Pak, which is a commonly available glucocorticoid taper that is administered over a short period of time after surgery. Our hypothesis is that the administration of the Medrol Dose Pak will lead to decreased pain, nausea, and opioid consumption in the weeks following total knee replacement.

DETAILED DESCRIPTION:
The study aims to evaluate the efficacy of a post-operative course of glucocorticoids on pain, range of motion, and extremity function after total knee replacement surgery. The goal is to compare the effects of a Medrol dose pak administration to the standard of care, which includes a single intraoperative dose of 10 mg intravenous dexamethasone, on postoperative outcomes. The study is important in the field because it aims to evaluate the effectiveness of glucocorticoids in reducing pain, nausea, and opioid consumption following total knee replacement surgery. The study will provide valuable insight into the role and optimal dosing of oral glucocorticoids after total knee replacement surgery (TKA). The results of this study could potentially improve postoperative outcomes for patients undergoing TKA. The study population in this randomized control trial consists of patients undergoing total knee replacement surgery. Patients will be randomly assigned to one of two treatment arms: (1) a single intraoperative dose of 10 mg intravenous dexamethasone (control group) or (2) a single intraoperative dose of 10 mg intravenous dexamethasone followed by a 6-day oral methylprednisolone taper course. The study does not mention any populations of increased concern. The study will last approximately 6 months with encounters at normal times within the clinic. The Emory r extremity surgeons will personally contact all patients for 1-day post-operation (standard of care for them) and at 7-10 days. Recruitment will occur at Emory University Orthopaedics & Spine Hospital. The study team will enroll 100 patients per group - 200 total.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total knee arthroplasty for osteoarthritis of the knee.
* Patients of the ages of 18 and 95 years.

Exclusion Criteria:

* Patients with concurrent and significant injuries to other bones or organs.
* Minors unable to consent for participation in the study.
* Subjects who, in the opinion of the investigator, may be non-compliant with study schedules or procedures.
* Patients with pre-existing immune suppression, where further immune suppression with glucocorticoids could warrant unwarranted or unneeded risk.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Score during Follow up period | Immediately after the surgery, day 1, day 2, day 3, day 4, day 5, day 6 and day 7 post-surgery
  A pain assessment will be assessed at each post-operative visit via the Visual Analog Pain Scale (VAS-pain), which is ranked from 0 (no pain) to 10 (highest amount of pain).
  Pain will be assessed at rest and during active movement of extremity. Patients will also be asked to fill out the VAS-pain score each day until post-op day 7.
Changes in Nausea score during Follow Up Period | Immediately after the surgery, day 1, day 2, day 3, day 4, day 5, day 6 and day 7 post-surgery
  : A nausea assessment will be assessed at each post-operative visit via the Visual Analog Nausea Scale (VAS-nausea), which is ranked from 0 (no nausea) to 10 (highest amount of nausea). Patients will be asked to fill out the VAS-nausea each day until post-operative day 7. Patients will also be monitored for post-operative vomiting.

SECONDARY OUTCOMES:
Changes in the postoperative range of motion following total knee arthroplasty (TKA) | Immediately before the surgery, Immediately after the surgery, day 1, day 2, day 3, day 4, day 5, day 6 and day 7 post-surgery
  Range of motion (ROM) assessment will take place at each clinic followed up with a hand-held goniometer. This will be done by assessing the total flexion-extension arc of the knee. ROM will be assessed as well in the preoperative holding area prior to surgery
Changes in post operative knee function utilizing Knee injury and Osteoarthritis Outcome Score (KOOS) | Day 1, day 2, day 3, day 4, day 5, day 6 and day 7 post-surgery
  The Patient-Related Knee Evaluation surveys. They have been used / validated in several studies and have a strong correlation with other scores. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems. These scores (and the KOOS, which the attending physician performs at follow up clinics after TKA) will be administered at each post-operative follow up.
Compare patient satisfaction with acute postoperative pain control | Immediately after the surgery, day 1, day 2, day 3, day 4, day 5, day 6 and day 7 post-surgery
  Patients will be asked about their pain control and satisfaction with the procedure and whether it meets or exceeds their expectations. The rating scale is much worse than expected, worse than expected, as expected, better than expected, or much better than expected.
Compare the postoperative opiate consumption measured as the number of tablets taken | Immediately after the surgery, day 1, day 2, day 3, day 4, day 5, day 6 and day 7 post-surgery
  Narcotic usage will be monitored, and the patient will be asked to count the amount of pain pills taken daily and this will be reported as part of the pain diary for the first 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Premkumar, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Musculoskeletal Institute, Atlanta, Georgia
  - Emory University Orthopaedics & Spine Hospital, Tucker, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT05859269/ICF_000.pdf